CLINICAL TRIAL: NCT06872099
Title: NAsal MEthicillin-resistant Staphylococcus (NAMES): a Prospective Study to Assess the Impact of Antibiotic Therapy on Nasal Colonization with Methicillin-resistant Staphylococcus Aureus (MRSA) in Hospitalized Children
Brief Title: NAsal MEthicillin-resistant Staphylococcus (NAMES): a Prospective Study to Assess the Impact of Antibiotic Therapy on Nasal Colonization with Methicillin-resistant Staphylococcus Aureus (MRSA) Inhospitalized Children
Acronym: NAMES
Status: Recruiting | Type: Observational
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Alessandra Ricciardi, MD, Fondazione IRCCS Policlinico San Matteo di Pavia
Other Study IDs: NAMES
Record Dates: First submitted 2025-03-06; First posted 2025-03-12 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: NAsal MEthicillin-resistant Staphylococcus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | US Export: No

SUMMARY:
Antimicrobial resistance (AMR) is recognized as one of the major threats to global health [1], causing up to 25.000 deaths in the European Union every year, longer hospitalizations and increased healthcare costs. It is well known that antimicrobial use is the main driving force towards AMR and up to 50% of antimicrobial prescriptions are either inappropriate or unnecessary [2]. It is then important to understand how to optimize antimicrobial usage not only in adults but also in infants, as they show different resistance patterns and have peculiar characteristics that may lead to incorrect administration and alteration of the pharmacokinetic and pharmacodynamic properties of the drug [3]. Antimicrobials are the most prescribed drugs in children [4][5] and this excessive usage has been recorded not only in developed countries, but also in low-income and middle-income ones [6]. In Europe, Italy reported one of the highest prescriptions rates, four times higher than the UK and six times higher than the Netherlands [7][8]. 84% of Italian infants in the community have already received at least one course of antibiotics at 2 years of age [9]. A point-prevalence survey (PPS) showed that 38.9% of hospitalized Italian infants received at least one antibiotic prescription both for treatment and prophylaxis; in children, the most commonly used antibiotic classes were third generation cephalosporins and penicillins plus enzyme inhibitors, with a high prescription rates of carbapenems and quinolones as well, often off-label [10]. In order to limit misuse and overuse of antibiotics in children, the joint SHEA-IDSA-PIDS position paper states the importance of introducing antimicrobial stewardship programs (ASPs) in all healthcare institutions [11].

Antimicrobial stewardship has been defined as "the optimal selection, dosage, and duration of antimicrobial therapy that results in the best clinical outcome for the treatment or prevention of infection, with minimal toxicity to the patient and minimal impact on subsequent resistance" [12]. So far, little progress has been made with developing pediatric ASPs, especially outside the United States healthcare system.

One of the most important studies conducted in Europe in this field, the ARPEC project, was designed as a PPS: this type of strategy is very useful if repeated regularly, as it allows to monitor prescription trends over time and to identify the problem of inappropriate antibiotic usage [13]. However, it has been shown that PPSs are not sufficient by themselves to change the clinical practice if not combined with other methods [14], such as pre-prescription authorization, prospective audit and feedback, educational and training programmes or technological means of support. In USA, methicillin-resistant Staphylococcus aureus (MRSA) in children mainly causes skin and soft tissue infections but invasive diseases were increasingly reported in 1995-2010 [15]. Studies on MRSA carriage in healthy children showed great geographic variation (from less than 1% in Belgium to 15% in Taiwan) that depend on many local differences [16]. Nevertheless, very few studies have been performed on the influence of antibiotic prescription in the acquisition of resistant microorganism such MRSA in pediatric population.

The aim of this study is to estimate the incidence of MRSA nasal colonization and invasive disease and to investigate the impact of antibiotic treatment during hospitalization on the acquisition of MRSA nasal colonization in children.

ELIGIBILITY:
Inclusion Criteria: · All the hospitalized children, aged between 1 and 16 years.

* Informed consent signed by parents or legal tutors

Exclusion Criteria: · All the hospitalized children admitted to the Unit of Oncologic/Hematologic disease or children affected with an hematologic disease also if admitted to the General Paediatric Ward.

* All the hospitalized children admitted to the Paediatric Intensive Care Unit (PICU)
* All the hospitalized children aged < 1 years old
* Children with parents or legal tutor who eventually refuse to sign the study consent form

Ages: 1 Year to 16 Years | Sex: All
Age Groups: Child
Study Population: The population enrolled in this study will include all the patients admitted to the Paediatric Unit of the involved Hospitals during the study period that respect inclusion and exclusion criteria
Sampling Method: Probability Sample
Enrollment: 76 (Estimated)
Dates: Start 2021-11-06 (Actual); Primary Completion 2025-02-19 (Actual); Study Completion 2025-03-19 (Estimated)

PRIMARY OUTCOMES:
Estimation of cumulative incidence of new MRSA nasal colonization in hospitalized pediatric patient. | 30 days

SECONDARY OUTCOMES:
Comparison of cumulative incidence of new MRSA nasal colonization between pediatric patients who received an antibiotic treatment and those who didn't receive it during hospitalization. | 30 days

OTHER OUTCOMES:
Estimation of cumulative incidence of MRSA invasive infection in hospitalized pediatric patient. | 30 days
Comparison of MRSA nasal colonization between different antibiotic classes' administration | 30 days
Estimation of the prevalence of MRSA colonization at the time of admission | 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Policlinico San Matteo, SC Malattie Infettive 1, Pavia, Pavia, Italy